CLINICAL TRIAL: NCT02951533
Title: Multicenter, Randomized, Open-Label, Efficacy Assessor-Blinded, Active Comparator-Controlled Phase 3b Study to Compare the Efficacy of Guselkumab to Fumaric Acid Esters (Fumaderm Initial/ Fumaderm) for Adult Patients With Moderate to Severe Plaque Psoriasis Who Are Candidates for and Naive to Systemic Treatment
Brief Title: A Study to Compare the Efficacy of Guselkumab to Fumaric Acid Esters for the Treatment of Participants With Moderate to Severe Plaque Psoriasis
Acronym: POLARIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag G.m.b.H (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108220; 2016-002135-15 (EudraCT Number); CNTO1959PSO3008 (Other: Janssen-Cilag G.m.b.H, Germany)
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — guselkumab; Fumarates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Group I: Guselkumab (Experimental): Participants will receive Guselkumab 100 milligram (mg) administered as 100 milligram per milliliter (mg/mL) solution subcutaneously (SC) by single-use prefilled syringe (PFS) at weeks 0, 4, 12 and 20.
  Interventions: Drug: Guselkumab
- Group II: Fumaric Acid Esters (FAE) (Active Comparator): Participants will receive Fumaderm initial/Fumaderm tablets by self administration at week 0. The individual FAE dose representing the optimal efficacy/tolerability ratio needs to be determined for each participant according to local prescription information. To this aim, FAE doses will be slowly increased beginning with increasing doses of Fumderm initial (containing 30 mg dimethylfumarate) over the first 3 weeks. Thereafter, participants will be switched to Fumaderm tablets (containing 120 mg dimethylfumarate) starting with 1 tablet per day. Fumaderm dose may be increased to a maximum of 3*2 tablets per day. The decision to maintain, increase or decrease the FAE dose depends on efficacy, safety and tolerability.
  Interventions: Drug: Fumaric Acid Esters

INTERVENTIONS:
Drug: Guselkumab — Participants will receive 100 mg of Guselkumab as 100 mg/mL solution subcutaneously.
  Arms: Group I: Guselkumab
Drug: Fumaric Acid Esters — Participants will receive Fumaderm initial/ Fumaderm tablets through self-administration.
  Arms: Group II: Fumaric Acid Esters (FAE)

SUMMARY:
The purpose of the study is to compare the efficacy of Guselkumab with commercially available active comparator Fumaderm initial/Fumaderm tablets for the treatment of adult participants with moderate to severe plaque-type psoriasis who have not yet received any systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of plaque-type psoriasis for at least 6 months before the first administration of study drug
* Have a Psoriasis Area and Severity Index (PASI) greater than (>)10 or Body Surface Area (BSA) >10 at screening and at baseline
* Have a Dermatology Life Quality Index (DLQI) >10 at screening and at baseline
* Agree not to receive a live virus or live bacterial vaccination during the study, or within 3 months after the last administration of study drug; for information on Bacille Calmette-Guérin (BCG) vaccination, agree not to receive a BCG vaccination during the study, or within 12 months after the last administration of study drug
* No dipstick detection of proteins or glucose in urine. If there are signs of proteins and/or glucose on urine test strip, the urine sample must be analyzed centrally. Here, protein and glucose levels must not exceed trace levels, example, <=(+); one re-test (central urine analysis) is allowed

Exclusion Criteria:

* Has a history or current signs or symptoms of severe, progressive, or uncontrolled liver or renal insufficiency, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Participants with nonplaque forms of psoriasis (for example, erythrodermic, guttate, or pustular) or with current drug-induced psoriasis (for example, a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium)
* Known allergies, hypersensitivity, or intolerance to Guselkumab or its excipients
* Is pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 12 weeks after the last dose of study drug
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (for example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2017-09-13 (Actual); Study Completion 2019-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag G.m.b.H, Germany Clinical Trial, Study Director — Janssen-Cilag G.m.b.H
Locations (28):
- Germany (28):
  - Augsburg
  - Berlin
  - Bielefeld
  - Dresden
  - Dülmen
  - Düsseldorf
  - Erlangen
  - Essen
  - Frankfurt
  - Gera
  - Hamburg
  - Heidelberg
  - Jena
  - Kiel
  - Leipzig
  - Lübeck
  - Mahlow
  - Mainz
  - Memmingen
  - München
  - Münster
  - Neu-Ulm
  - Osnabrück
  - Selters
  - Stuttgart
  - Tübingen
  - Witten
  - Wuppertal

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total of 119 participants were enrolled and randomized, 118 (GUS [60], FAE [58 participants]) were treated in this study. Out of them, 42 participants completed study in Part III.
Groups:
- Guselkumab (GUS): Participants received guselkumab (GUS) 100 milligram (mg) administered as 100 mg per milliliter (mg/mL) solution subcutaneously (SC) at Weeks 0, 4, then every 8 weeks (at Week 12 and 20 - Part I). Participants who completed Part I continued to receive GUS 100 mg at Week 28 and 32 - Part IIa. At Week 32, PASI 75 response was evaluated. PASI 75 responders and non-responders of GUS arm continued to receive GUS 100 mg SC every 8 weeks (Weeks 36, 44 and 52). PASI 75 non-responders of FAE switched to 100 mg GUS SC at Week 32, continued at Week 36, 44 and 52 (Part IIb). Safety follow-up was done at Week 32 (Part I), Week 64 (Part II) and up to 12 weeks after discontinuing drug. Participants who received GUS in Part II (who started GUS at Week 0/ switched from FAE to GUS at Week 32), had no psoriatic arthritis at baseline and achieved PASI 90 response at end of Part II (Week 56), entered follow-up extension at Week 64 in Part III and followed-up until loss of response/ until Week 100.
- Fumaric Acid Esters (FAE): Participants received FAE tablets by self-administration at Week 0. Doses were up-titrated and were taken every day with different daily doses depending on optimal individual benefit risk ratio (maximum 6*120 mg/day) as per local prescribing information up to Week 24 (Part I). Participants who completed Part I and consented for Part IIa continued to receive same treatment up to Week 32 (Part IIa). At Week 32, PASI 75 response was evaluated and PASI 75 responders of FAE arm continued to receive commercially available FAE tablets specifically labeled for study (Part IIb) up to Week 56. PASI 75 non-responders of FAE arm switched to 100 mg GUS at Week 32 and received 100 mg GUS SC at Week 36, 44 and Week 52 (Part IIb). For participants who discontinued study, safety follow-up was done at Week 32 (Part I) / Week 64 (Part II) or 12 weeks after last treatment (whatever came first). For all participants who continued study, safety was followed-up at every visit.
- FAE to Guselkumab: At Week 32, PASI 75 response was evaluated and PASI 75 non-responders of FAE arm were switched to GUS and received GUS 100 mg SC at Weeks 32, 36, 44 and 52. Safety follow-up was done at Week 64 (Part II). Participants who discontinued at any timepoint were followed-up 12 weeks after last treatment dose. Participants who received GUS in Study Part II (participants who switched from FAE to GUS treatment at Week 32), had no psoriatic arthritis at baseline and achieved a PASI 90 response at end of Study Part II (Week 56) entered follow-up extension at Week 64 in Study Part III (GUS withdrawal phase) and were followed-up until loss of response or until Week 100.
Period: Part I (Week 0 Through Week 24)
Arm/Group | Guselkumab (GUS) | Fumaric Acid Esters (FAE) | FAE to Guselkumab
Started | 60 | 59 | 0
Treated | 60 | 58 | 0
Completed | 56 | 36 | 0
Not Completed | 4 | 23 | 0
Not completed — Adverse Event | 0 | 16 | 0
Not completed — Lost to Follow-up | 2 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 0
Not completed — Noncompliance with Study Drug | 0 | 1 | 0
Period: Part IIa (Week 24 Through Week 32)
Arm/Group | Guselkumab (GUS) | Fumaric Acid Esters (FAE) | FAE to Guselkumab
Started | 56 | 35 (1 participant did not sign informed consent form (ICF) for Study Part II but completed Study Part I.) | 0
PASI 75 Responder at Week 32 | 54 | 14 | 0
PASI 75 Non-responder at Week 32 | 1 | 20 | 0
Completed | 55 | 34 | 0
Not Completed | 1 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Part IIb (Week 32 Through Week 56)
Arm/Group | Guselkumab (GUS) | Fumaric Acid Esters (FAE) | FAE to Guselkumab
Started | 55 | 14 (Out of 34 participants in the FAE group, 14 PASI 75 responders remained on FAE treatment.) | 20 (Out of 34 participants in FAE group, 20 PASI 75 non-responders switched to GUS group.)
Completed | 54 | 10 | 20
Not Completed | 1 | 4 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0
Period: Part III (Week 64 Through Week 100)
Arm/Group | Guselkumab (GUS) | Fumaric Acid Esters (FAE) | FAE to Guselkumab
Started | 36 (18 participants were not eligible to enter Part III.) | 0 (10 participants in the FAE group were not eligible to enter Part III.) | 12 (8 participants were not eligible to enter Part III.)
Completed | 32 | 0 | 10
Not Completed | 4 | 0 | 2
Not completed — Prohibited Medication Therapy | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Guselkumab (GUS) | Fumaric Acid Esters (FAE) | Total
Number analyzed (Participants) | 60 | 59 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (13.98) | 45.8 (13.72) | 42.4 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 40 | 42 | 82
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 57 | 57 | 114
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 60 | 59 | 119

OUTCOME MEASURES:

1. Primary Outcome: Part I: Percentage of Participants Who Achieved Psoriasis Area and Severity Index (PASI) 90 Response at Week 24
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percent [%] to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produces a numeric score that can range from 0 (no visible skin involvement) to 72 (maximal skin involvement of the whole body). A higher score indicates more severe disease. A PASI 90 response represents participants who achieved at least a 90 % improvement from baseline in the PASI score.
Time Frame: At Week 24
Population: Efficacy analysis set (EAS) included all participants who were randomized to one of the two treatment groups (GUS or FAE) at Week 0 regardless of the treatment they actually received. Missing data was imputed using non-responder imputation (NRI) (participants with missing data at Week 4,16 and 24 were considered non-responders).
Measure: Number; unit: Percentage of Participants
Groups:
- Part I: Guselkumab (GUS): Participants received GUS 100 milligram (mg) treatment administered as 100 milligram per milliliter (mg/mL) solution subcutaneously (SC) at Weeks 0, 4, 12 and 20. Participants who completed the treatment phase until Week 24 entered the Part II of the study.
- Part I: Fumaric Acid Esters (FAE): Participants received FAE initial/FAE tablets by self-administration at Week 0. The doses were uptitrated and had to be taken every day with different daily doses depending on the optimal individual benefit risk ratio (maximum 6*120 mg/day) according to local prescribing information up to Week 24. Participants who completed the treatment phase until Week 24 entered the Part II of the study.
Arm/Group | Part I: Guselkumab (GUS) | Part I: Fumaric Acid Esters (FAE)
Number analyzed (Participants) | 60 | 59
Percentage of Participants | 81.7 | 13.6
Statistical Analysis 1: Comparison: Part I: Guselkumab (GUS) vs Part I: Fumaric Acid Esters (FAE); Test type: Superiority; p < 0.0001, Chi-squared

2. Secondary Outcome: Part I: Percentage of Participants Who Achieved PASI 75 Response at Week 24
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percent [%] to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produces a numeric score that can range from 0 (no visible skin involvement) to 72 (maximal skin involvement of the whole body). A higher score indicates more severe disease. A PASI 75 response represents participants who achieved at least a 75 % improvement from baseline in the PASI score.
Time Frame: At Week 24
Population: EAS included all participants who were randomized to one of the two treatment groups (GUS or FAE) at Week 0 regardless of the treatment they actually received. Missing data was imputed using NRI (participants with missing data at Week 4,16 and 24 were considered non-responders).
Measure: Number; unit: Percentage of Participants
Arm/Group | Part I: Guselkumab (GUS) | Part I: Fumaric Acid Esters (FAE)
Number analyzed (Participants) | 60 | 59
Percentage of Participants | 90.0 | 27.1

3. Secondary Outcome: Part I: Percentage of Participants Who Achieved a Dermatology Life Quality Index (DLQI) Score of Less Than or Equal to (=<) 1 at Week 24
Description: The DLQI is a 10-item questionnaire that measures the impact of skin disease on participant's quality of life, can be used to assess 6 different aspects that may affect quality of life 1) symptoms and feelings, 2) daily activities, 3) leisure, 4) work or school performance, 5) personal relationships, and 6) treatment. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicate more impact on quality of life. The DLQI produces a total numeric score that can range from 0 (not at all) to 30 (very much): 0-1 = no effect at all on the participant's life; 2-6 = small effect on the participant's life; 7-12 = moderate effect on the participant's life; 13-18 = very large effect on the participant's life; 19-30 = extremely large effect on the participant's life. A higher score indicates a low quality of life due to more severe disease.
Time Frame: At Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Part I: Guselkumab (GUS) | Part I: Fumaric Acid Esters (FAE)
Number analyzed (Participants) | 60 | 59
Percentage of Participants | 61.7 | 16.9

4. Secondary Outcome: Part I: Percentage of Participants Who Achieved PASI 100 Response at Week 24
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percent [%] to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produces a numeric score that can range from 0 (no visible skin involvement) to 72 (maximal skin involvement of the whole body). A higher score indicates more severe disease. A PASI 100 response represents participants who achieved a 100% improvement from baseline in the PASI score.
Time Frame: At Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Part I: Guselkumab (GUS) | Part I: Fumaric Acid Esters (FAE)
Number analyzed (Participants) | 60 | 59
Percentage of Participants | 31.7 | 3.4

5. Secondary Outcome: Part I: Change From Baseline in the Signs and Symptoms Aggregate Scores of the Psoriasis Symptoms and Signs Diary (PSSD) Score at Week 24
Description: The PSSD (7-day version) is a patient-reported outcome (PRO) questionnaire designed and validated to measure the severity of psoriasis symptoms and signs for the assessment of treatment benefit. It consisted of 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 (absent) to 10 (worst imaginable) numerical rating scales for severity. Items were averaged on the daily symptom score and sign score when at least 3 items greater than or equal to (>=) 50 percentage of 5 items on these scales are answered. The average value is converted into 0-100 scoring, such that Symptom [or Sign] score=average value*10, where, 0= least severe and 100=most severe and higher score indicates more severe disease.
Time Frame: Baseline and Week 24
Population: EAS included all participants who were randomized to one of two treatment groups (GUS or FAE) at Week 0 regardless of treatment they received. Missing data was imputed using last observed carried forward (LOCF) imputation method. Here N (number of participants analyzed) signifies number of participants evaluable for this outcome measure (OM).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part I: Guselkumab (GUS) | Part I: Fumaric Acid Esters (FAE)
Number analyzed (Participants) | 60 | 58
Units on a scale
  Sign score | -59.8 (18.3) | -39.7 (26.7)
  Symptom score | -52.0 (22.0) | -34.0 (25.4)

6. Secondary Outcome: Part I: Change From Baseline in the Individual Scale Scores for Itch, Pain, and Scaling of PSSD Components at Week 24
Description: The PSSD (7 day version) is a patient-reported outcome (PRO) questionnaire designed and validated to measure the severity of psoriasis symptoms and signs for the assessment of treatment benefit. It consisted of 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 (absent) to 10 (worst imaginable) numerical rating scales for severity. Items were averaged on the daily symptom score and sign score when at least 3 items (>=50 percentage of 5 items) on these scales are answered. The average value is converted into 0-100 scoring, such that Symptom [or Sign] score = average value*10, where, 0= least severe and 100= most severe and higher score indicates more severe disease.
Time Frame: Baseline and Week 24
Population: EAS included all participants who were randomized to one of the two treatment groups (GUS or FAE) at Week 0 regardless of the treatment they received. Missing data was imputed using LOCF imputation method. Here N (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part I: Guselkumab (GUS) | Part I: Fumaric Acid Esters (FAE)
Number analyzed (Participants) | 60 | 58
Units on a scale
  Itch score | -5.85 (2.83) | -3.90 (2.86)
  Pain score | -5.07 (2.86) | -2.93 (3.12)
  Scaling score | -6.48 (2.25) | -4.43 (3.02)

7. Secondary Outcome: Part I: Percentage of Participants Who Achieved an Absolute PASI Score Less Than or Equal to (=<) 1 at Week 24
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percent [%] to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produces a numeric score that can range from 0 (no visible skin involvement) to 72 (maximal skin involvement of the whole body). A higher score indicates more severe disease. Percentage of Participants who Achieved an absolute PASI score less than or equal to (=<) 1 were assessed.
Time Frame: At Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Part I: Guselkumab (GUS) | Part I: Fumaric Acid Esters (FAE)
Number analyzed (Participants) | 60 | 59
Percentage of Participants | 66.7 | 10.2

8. Secondary Outcome: Part I: Percentage of Participants Who Achieved an Investigator's Global Assessment (IGA) Score 0 at Week 24
Description: The Investigator's Global Assessment (IGA) documents the investigator's assessment of the participant's psoriasis at a given time. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Time Frame: At Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Part I: Guselkumab (GUS) | Part I: Fumaric Acid Esters (FAE)
Number analyzed (Participants) | 60 | 59
Percentage of Participants | 51.7 | 6.8

9. Secondary Outcome: Part I: Change From Baseline in Percent Body Surface Area (%BSA) Psoriatic Involvement at Week 24
Description: BSA as physical measure to define disease severity is to determine how much of the Body Surface Area (BSA) is affected by psoriasis. Involved BSA is calculated by using the palm of the participant's hand as equivalent to 1% of the BSA (rule of palm). Psoriasis affected BSA under 5% suggests mild psoriasis, a BSA of 5% to 10% is considered moderate, and an involved BSA of over 10% indicates severe psoriasis.
Time Frame: Baseline and Week 24
Population: EAS included all participants who were randomized to one of the two treatment groups (GUS or FAE) at Week 0 regardless of the treatment they actually received. Missing data was imputed using LOCF imputation method. Here "N" (Number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Change in BSA (% points)
Arm/Group | Part I: Guselkumab (GUS) | Part I: Fumaric Acid Esters (FAE)
Number analyzed (Participants) | 59 | 57
Change in BSA (% points) | -18.5 (10.4) | -9.2 (11.2)

10. Secondary Outcome: Part I: Change From Baseline in DLQI Score at Week 24
Description: as for outcome 3
Time Frame: Baseline and Week 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part I: Guselkumab (GUS) | Part I: Fumaric Acid Esters (FAE)
Number analyzed (Participants) | 60 | 58
Units on a scale | -15.2 (5.1) | -9.4 (7.2)

11. Secondary Outcome: Part I: Percentage of Participants Who Achieved an Scalp Specific Investigator´s Global Assessment (Ss-IGA) Score of Absence of Disease (0) at Week 24
Description: The ss-IGA instrument is used to evaluate the disease severity of scalp psoriasis (SP). The lesions are assessed in terms of the clinical signs of redness, thickness, and scaliness which are scored as: absence of disease (0), very mild disease (1), mild disease (2), moderate disease (3), and severe disease (4).
Time Frame: At Week 24
Population: EAS: participants randomized to one of two treatments (GUS or FAE) at Week 0 regardless of treatment received and SP, ss-IGA Score>=2 at Baseline. Missing data was imputed using NRI (participants with missing data at Week 4,16, 24 were non-responders).
Measure: Number; unit: Percentage of Participants
Arm/Group | Part I: Guselkumab (GUS) | Part I: Fumaric Acid Esters (FAE)
Number analyzed (Participants) | 54 | 53
Percentage of Participants | 48.1 | 13.2

12. Secondary Outcome: Part I: Change From Baseline in 36-Item Short-Form Health Survey Version 2 (SF-36 V2) Physical Component Summary (PCS) and Mental Component Summary (MCS) at Week 24
Description: SF-36 V2 is a generic 36-item questionnaire measuring health-related quality of life (HRQL) covering 2 summary measures: physical component summary (PCS) and mental component summary (MCS). The SF-36 consists of 8 subscales (physical function, role limitations due to physical problems, pain, general health perception, vitality, social function, role limitations due to emotional problems, and mental health). Participants self-report on items in a subscale that have between 2-6 choices per item using Likert-type responses (e.g. none of the time, some of the time, etc.). Summations of item scores of the same subscale give the subscale scores, which are transformed into a range from 0 to 100; zero= worst HRQL, 100=best HRQL. Higher scores indicate better health status.
Time Frame: Baseline and Week 24
Population: EAS included all participants who were randomized to one of the two treatment groups (GUS or FAE) at Week 0 regardless of the treatment they received. Missing data was imputed using LOCF. Here "N" (Number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part I: Guselkumab (GUS) | Part I: Fumaric Acid Esters (FAE)
Number analyzed (Participants) | 59 | 57
Units on a scale
  SF-36 PCS scores | 8.0 (6.9) | 2.3 (8.2)
  SF-36 MCS scores | 5.8 (10.6) | 6.5 (9.3)

13. Secondary Outcome: Part IIb: Percentage of Participants With a PASI 75 Response at Week 32 Who Maintained Response at Week 56
Description: as for outcome 2
Time Frame: Week 56
Population: Study Part IIb analysis set included all participants who entered Study Part IIb and were treated with one of the two treatments (GUS or FAE) at least once during the treatment period from Week 32 to Week 56. Missing data was imputed using NRI (participants with missing data at Week 40, 48, and 56 were considered non-responders).
Measure: Number; unit: Percentage of Participants
Groups:
- Part IIb: Guselkumab (GUS): At Week 32 (study Part IIb), PASI 75 response was evaluated and PASI 75 responders and non-responders of GUS arm continued to receive GUS 100 mg SC every 8 weeks (Weeks 36, 44 and 52). For participants, who discontinued study, a safety follow-up was done at Week 64 (Part II)or 12 weeks after last treatment (whatever came first). For all participants who continued study, safety was followed-up at every visit.
- Part IIb: Fumaric Acid Esters (FAE): At Week 32, PASI 75 response was evaluated and PASI 75 responders of FAE arm continued to receive commercially available FAE tablets specifically labeled for the study (study Part IIb) up to Week 56. For participants, who discontinued study, a safety follow up was done at Week 64 (Part II)or 12 weeks after last treatment (whatever came first). For all participants who continued study, safety was followed-up at every visit.
Arm/Group | Part IIb: Guselkumab (GUS) | Part IIb: Fumaric Acid Esters (FAE)
Number analyzed (Participants) | 54 | 14
Percentage of Participants | 98.1 | 64.3

14. Secondary Outcome: Part IIb: Percentage of Participants With a PASI 90 Response at Week 32 Who Maintained Response at Week 56
Description: as for outcome 1
Time Frame: Week 56
Population: Study Part IIb analysis set included all participants who entered Study Part IIb and were treated with one of the two treatments (GUS or FAE) at least once during the treatment period from Week 32 to Week 56. Missing data was imputed using NRI (participants with missing data at Week 40,48 and 56 were considered non-responders).
Measure: Number; unit: Percentage of Participants
Arm/Group | Part IIb: Guselkumab (GUS) | Part IIb: Fumaric Acid Esters (FAE)
Number analyzed (Participants) | 54 | 14
Percentage of Participants | 85.2 | 35.7

15. Secondary Outcome: Part IIb: Percentage of Participants With DLQI Score of 0 or 1 at Week 32 Who Maintained Response at Week 56
Description: as for outcome 3
Time Frame: Week 56
Population: as for outcome 14
Measure: Number; unit: Percentage of Participants
Arm/Group | Part IIb: Guselkumab (GUS) | Part IIb: Fumaric Acid Esters (FAE)
Number analyzed (Participants) | 54 | 14
Percentage of Participants | 64.8 | 21.4

16. Secondary Outcome: Part IIb: Percentage of Participants With a PASI 75 Response at Week 56
Description: as for outcome 2
Time Frame: Week 56
Population: as for outcome 13
Measure: Number; unit: Percentage of Participants
Arm/Group | Part IIb: Guselkumab (GUS) | Part IIb: Fumaric Acid Esters (FAE)
Number analyzed (Participants) | 54 | 14
Percentage of Participants | 98.1 | 64.3

17. Secondary Outcome: Part IIb: Percentage of Participants With a PASI 90 Response at Week 56
Description: as for outcome 1
Time Frame: Week 56
Population: as for outcome 14
Measure: Number; unit: Percentage of Participants
Arm/Group | Part IIb: Guselkumab (GUS) | Part IIb: Fumaric Acid Esters (FAE)
Number analyzed (Participants) | 54 | 14
Percentage of Participants | 90.7 | 50.0

18. Secondary Outcome: Part IIb: Percentage of Participants With a PASI 100 Response at Week 56
Description: as for outcome 4
Time Frame: Week 56
Population: as for outcome 14
Measure: Number; unit: Percentage of Participants
Arm/Group | Part IIb: Guselkumab (GUS) | Part IIb: Fumaric Acid Esters (FAE)
Number analyzed (Participants) | 54 | 14
Percentage of Participants | 53.7 | 21.4

19. Secondary Outcome: Part IIb: Percentage of Participants With a DLQI Score of 0 or 1 at Week 56
Description: as for outcome 3
Time Frame: Week 56
Population: as for outcome 14
Measure: Number; unit: Percentage of Participants
Arm/Group | Part IIb: Guselkumab (GUS) | Part IIb: Fumaric Acid Esters (FAE)
Number analyzed (Participants) | 54 | 14
Percentage of Participants | 72.2 | 28.6

20. Secondary Outcome: Part I/IIa: Percentage of Participants Who Achieved PASI 75 Response at Week 32
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percent [%] to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produces a numeric score that can range from 0 (no visible skin involvement) to 72 (maximal skin involvement of the whole body). A higher score indicates more severe disease. A PASI 75 response represents participants who achieved at least a 75 % improvement from baseline in the PASI score. Data reported collectively for Part I and Part IIa (that is from Week 0 to Week 32) per planned analysis for this outcome measure (OM).
Time Frame: Week 32
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Groups:
- Part I/IIa: Guselkumab (GUS): In Part I, participants received GUS 100 mg treatment administered as 100 mg/mL solution SC at Weeks 0, 4, 12 and 20. Participants who completed treatment phase until Week 24 entered Part II of study. Participants who completed Part I continued to receive GUS 100 mg SC at Week 28 and 32 during study Part IIa. For participants who discontinued study, a safety follow-up was done at Week 32 (Part I) or 12 weeks after last treatment (whatever came first). For all participants who continued study, safety was followed-up at every visit.
- Part I/IIa: FAE: In Part I, participants received FAE tablets by self-administration at Week 0. The doses were up-titrated and had to be taken every day with different daily doses depending on the optimal individual benefit risk ratio (maximum 6*120 mg/day) according to local prescribing information up to Week 24. Participants who completed the treatment phase until Week 24 entered the Part II of the study. Participants who completed Part I and consented for Part IIa continued to receive commercially available FAE tablets specifically labeled for the study from Week 24 through Week 32 during study Part IIa. For participants who discontinued study, a safety follow-up was done at Week 32 (Part I) or 12 weeks after last treatment (whatever came first). For all participants who continued study, safety was followed-up at every visit.
Arm/Group | Part I/IIa: Guselkumab (GUS) | Part I/IIa: FAE
Number analyzed (Participants) | 60 | 59
Percentage of Participants | 90.0 | 23.7

21. Secondary Outcome: Part I/IIa: Percentage of Participants Who Achieved PASI 90 Response at Week 32
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percent [%] to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produces a numeric score that can range from 0 (no visible skin involvement) to 72 (maximal skin involvement of the whole body). A higher score indicates more severe disease. A PASI 90 response represents participants who achieved at least a 90 % improvement from baseline in the PASI score. Data reported collectively for Part I and Part IIa (that is from Week 0 to Week 32) per planned analysis for this OM.
Time Frame: Week 32
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Part I/IIa: Guselkumab (GUS) | Part I/IIa: FAE
Number analyzed (Participants) | 60 | 59
Percentage of Participants | 78.3 | 11.9

22. Secondary Outcome: Part I/IIa: Percentage of Participants Who Achieved PASI 100 Response at Week 32
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percent [%] to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produces a numeric score that can range from 0 (no visible skin involvement) to 72 (maximal skin involvement of the whole body). A higher score indicates more severe disease. A PASI 100 response represents participants who achieved a 100% improvement from baseline in the PASI score. Data reported collectively for Part I and Part IIa (that is from Week 0 to Week 32) per planned analysis for this OM.
Time Frame: Week 32
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Part I/IIa: Guselkumab (GUS) | Part I/IIa: FAE
Number analyzed (Participants) | 60 | 59
Percentage of Participants | 43.3 | 6.8

23. Secondary Outcome: Part I/IIa: Percentage of Participants With a DLQI Score of 0 or 1 at Week 32
Description: DLQI is 10-item questionnaire that measures impact of skin disease on participant's quality of life, can be used to assess 6 different aspects that may affect quality of life 1) symptoms and feelings, 2) daily activities, 3) leisure, 4) work or school performance, 5) personal relationships, and 6) treatment. Each question was evaluated on 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicate more impact on quality of life. DLQI produces total numeric score ranging from 0 (not at all) to 30 (very much): 0-1=no effect at all on participant's life; 2-6 =small effect on participant's life; 7-12 = moderate effect on participant's life; 13-18 =very large effect on participant's life; 19-30 =extremely large effect on participant's life. Higher score indicates low quality of life due to more severe disease. Data reported collectively for Part I and Part IIa (that is from Week 0 to Week 32) per planned analysis for this OM.
Time Frame: Week 32
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Part I/IIa: Guselkumab (GUS) | Part I/IIa: FAE
Number analyzed (Participants) | 60 | 59
Percentage of Participants | 63.3 | 16.9

24. Secondary Outcome: Part III: Percentage of Participants With a PASI 90 Response at Week 56 Who Maintained Response (That is Who Had PASI Score <=5) at Week 100 After Drug Withdrawal
Description: as for outcome 1
Time Frame: Week 100
Population: Study Part III analysis set included all participants who were treated with GUS during Part IIb (Weeks 32 to 64 of Study, and who were withdrawn from study treatment) and entered Part III. Missing data was imputed using NRI (participants with missing data at Week 64,76,88 and 100 were non-responders).
Measure: Number; unit: Percentage of Participants
Groups:
- Part III: Guselkumab (GUS): Participants who received guselkumab in Study Part II (participants who started guselkumab treatment at Week 0), had no psoriatic arthritis diagnosed at baseline and achieved a PASI 90 response at end of Study Part II (Week 56) entered follow-up extension at Week 64 in Study Part III (GUS withdrawal phase) and were followed-up until loss of response or until Week 100 at the latest.
- Part III: FAE to Guselkumab: At Week 32, PASI 75 response was evaluated and PASI 75 non-responders of FAE arm were switched to GUS and received GUS 100 mg SC at Week 32, 36, 44 and 52. Safety follow-up was done at Week 64 (Part II). Participants who discontinued at any timepoint were followed-up 12 weeks after last treatment dose. Participants who switched from FAE to GUS treatment at Week 32, had no psoriatic arthritis at baseline and achieved a PASI 90 response at end of Study Part II (Week 56) entered follow-up extension at Week 64 in Study Part III (GUS withdrawal phase) and were followed-up until loss of response or until Week 100.
Arm/Group | Part III: Guselkumab (GUS) | Part III: FAE to Guselkumab
Number analyzed (Participants) | 36 | 12
Percentage of Participants | 47.2 | 25.0

25. Secondary Outcome: Part III: Time to Loss of Response (PASI >5) From Week 56 After Guselkumab Withdrawal at Week 100
Description: The time to loss of response from Week 56 after guselkumab withdrawal at Week 100 was calculated as time from Week 56 to first onset of loss of response (PASI >5). The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percent [%] to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produces a numeric score that can range from 0 (no visible skin involvement) to 72 (maximal skin involvement of the whole body). A higher score indicates more severe disease.
Time Frame: Week 100
Population: Study Part III analysis set included all participants who were treated with guselkumab during Study Part IIb (Weeks 32 to 64 of the Study, and who were withdrawn from study treatment) and entered Study Part III. Results were reported for observed cases.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part III: Guselkumab (GUS) | Part III: FAE to Guselkumab
Number analyzed (Participants) | 36 | 12
Days | 315 [301 to NA] — The upper bound of the 95 percent confidence interval (CI) for median was not reached due to insufficient event rate. | 293 [219 to 315]

26. Secondary Outcome: Part III: Time to PASI >3 From Week 56 After Guselkumab Withdrawal at Week 100
Description: The time to PASI>3 from Week 56 after guselkumab withdrawal at Week 100 was calculated as time from Week 56 to PASI response that is PASI >3. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percent [%] to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produces a numeric score that can range from 0 (no visible skin involvement) to 72 (maximal skin involvement of the whole body). A higher score indicates more severe disease.
Time Frame: Week 100
Population: as for outcome 25
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part III: Guselkumab (GUS) | Part III: FAE to Guselkumab
Number analyzed (Participants) | 36 | 12
Days | 306 [227 to 308] | 226 [141 to 308]

27. Secondary Outcome: Part III: Time to Loss of Response (PASI >5) From Week 52 After Guselkumab Withdrawal at Week 100
Description: The time to loss of response from Week 52 after guselkumab withdrawal at Week 100 was calculated as time from Week 52 to first onset of loss of response (PASI >5). The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percent [%] to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produces a numeric score that can range from 0 (no visible skin involvement) to 72 (maximal skin involvement of the whole body). A higher score indicates more severe disease.
Time Frame: Week 100
Population: as for outcome 25
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part III: Guselkumab (GUS) | Part III: FAE to Guselkumab
Number analyzed (Participants) | 36 | 12
Days | 336 [322 to NA] — The upper bound of the 95 percent confidence interval (CI) for median was not reached due to insufficient event rate. | 321 [251 to 350]

28. Secondary Outcome: Part III: Time to PASI >3 From Week 52 After Guselkumab Withdrawal at Week 100
Description: The time to PASI>3 from Week 52 after guselkumab withdrawal at Week 100 was calculated as time from Week 52 to PASI response that is PASI >3. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percent [%] to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produces a numeric score that can range from 0 (no visible skin involvement) to 72 (maximal skin involvement of the whole body). A higher score indicates more severe disease.
Time Frame: Week 100
Population: as for outcome 25
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part III: Guselkumab (GUS) | Part III: FAE to Guselkumab
Number analyzed (Participants) | 36 | 12
Days | 334 [252 to 337] | 254 [173 to 329]

29. Secondary Outcome: Part III: Percentage of Participants With PASI 90 Response at Week 56 Who Maintained PASI 90 Response at Week 100 After Drug Withdrawal
Description: as for outcome 1
Time Frame: Week 100
Population: Study Part III analysis set included all participants who were treated with guselkumab during Study Part IIb (Weeks 32 to 64 of the Study, and who were withdrawn from study treatment) and entered Study Part III. Missing data was imputed using NRI (participants with missing data at Week 64,76,88 and 100 were considered non-responders).
Measure: Number; unit: Percentage of Participants
Arm/Group | Part III: Guselkumab (GUS) | Part III: FAE to Guselkumab
Number analyzed (Participants) | 36 | 12
Percentage of Participants | 13.9 | 8.3

30. Secondary Outcome: Part III: Percentage of Participants Who Achieved PASI 100 Response at Week 100
Description: as for outcome 4
Time Frame: Week 100
Population: as for outcome 29
Measure: Number; unit: Percentage of Participants
Arm/Group | Part III: Guselkumab (GUS) | Part III: FAE to Guselkumab
Number analyzed (Participants) | 36 | 12
Percentage of Participants | 5.6 | 0.0

31. Secondary Outcome: Part III: Percentage of Participants Who Achieved an Absolute PASI Score <=1, <=2, <=3, <=5 at Week 100
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percent [%] to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produces a numeric score that can range from 0 (no visible skin involvement) to 72 (maximal skin involvement of the whole body). A higher score indicates more severe disease.
Time Frame: Week 100
Population: as for outcome 24
Measure: Number; unit: Percentage of Participants
Arm/Group | Part III: Guselkumab (GUS) | Part III: FAE to Guselkumab
Number analyzed (Participants) | 36 | 12
Percentage of Participants
  PASI Score <=1 | 8.3 | 0.0
  PASI Score <=2 | 19.4 | 8.3
  PASI Score <=3 | 30.6 | 16.7
  PASI Score <=5 | 47.2 | 25.0

32. Secondary Outcome: Part III: Change From Baseline (Week 56) in Signs and Symptoms Aggregate Scores of the Psoriasis Symptom and Sign Diary (PSSD) Total Score at Week 100
Description: as for outcome 5
Time Frame: Baseline (Week 56) and Week 100
Population: Study Part III analysis set included all participants who were treated with guselkumab during Study Part IIb (Weeks 32 to 64 of the Study, and who were withdrawn from study treatment) and entered Study Part III. Missing data was imputed using last observed carried forward (LOCF) imputation method.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part III: Guselkumab (GUS) | Part III: FAE to Guselkumab
Number analyzed (Participants) | 36 | 12
Units on a scale
  Symptom Score at Baseline (Week 56) | 3.4 (5.4) | 11.2 (13.2)
  Change in Symptom score at Week 100 | 25.1 (24.7) | 30.7 (21.7)
  Sign Score at Baseline (Week 56) | 5.4 (9.3) | 13.5 (12.9)
  Change in Sign score at Week 100 | 29.4 (24.8) | 37.9 (28.7)

33. Secondary Outcome: Part III: Percentage of Participants Who Achieved an Investigator's Global Assessment (IGA) Score of 0 at Week 100
Description: as for outcome 8
Time Frame: Week 100
Population: Study Part III analysis set included all participants who were treated with guselkumab during Study Part IIb (Weeks 32 to 64 of the Study, and who were withdrawn from study treatment) and entered Study Part III. Missing data was imputed using NRI (participants with missing data at Week 64, 76,88 and 100 were considered non-responders).
Measure: Number; unit: Percentage of participants
Arm/Group | Part III: Guselkumab (GUS) | Part III: FAE to Guselkumab
Number analyzed (Participants) | 36 | 12
Percentage of participants | 8.3 | 0.0

34. Secondary Outcome: Part III: Percentage of Participants Who Achieved an Investigator's Global Assessment (IGA) Score of 0 or 1 at Week 100
Description: as for outcome 8
Time Frame: Week 100
Population: as for outcome 33
Measure: Number; unit: Percentage of participants
Arm/Group | Part III: Guselkumab (GUS) | Part III: FAE to Guselkumab
Number analyzed (Participants) | 36 | 12
Percentage of participants | 30.6 | 16.7

35. Secondary Outcome: Part III: Change From Baseline (Week 56) in Percent Body Surface Area (%BSA) Psoriatic Involvement at Week 100
Description: as for outcome 9
Time Frame: Baseline (Week 56) and Week 100
Population: Study Part III analysis set included all participants who were treated with guselkumab during Study Part IIb (Weeks 32 to 64 of the Study, and who were withdrawn from study treatment) and entered Study Part III. Missing data was imputed using LOCF imputation method.
Measure: Mean (Standard Deviation); unit: Change in BSA (% points)
Arm/Group | Part III: Guselkumab (GUS) | Part III: FAE to Guselkumab
Number analyzed (Participants) | 36 | 12
Change in BSA (% points)
  Baseline (Week 56) | 0.9 (1.2) | 1.5 (2.1)
  Change at Week 100 | 6.1 (6.3) | 9.1 (5.8)

36. Secondary Outcome: Part III: Percentage of Participants With a DLQI Score of 0 or 1 at Week 100
Description: as for outcome 3
Time Frame: Week 100
Population: as for outcome 35
Measure: Number; unit: Percentage of participants
Arm/Group | Part III: Guselkumab (GUS) | Part III: FAE to Guselkumab
Number analyzed (Participants) | 36 | 12
Percentage of participants | 25 | 8.3

37. Secondary Outcome: Part III: Change From Baseline in DLQI Score at Week 100
Description: as for outcome 3
Time Frame: Baseline (Week 56) and Week 100
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part III: Guselkumab (GUS) | Part III: FAE to Guselkumab
Number analyzed (Participants) | 36 | 12
Units on a scale
  Baseline (Week 56) | 0.9 (1.3) | 3.5 (4.0)
  Change at Week 100 | 5.3 (6.0) | 8.0 (5.4)

38. Secondary Outcome: Part III: Percentage of Participants With a DLQI Score of 0 or 1 at Week 56 Who Maintained Response at Week 100
Description: as for outcome 3
Time Frame: Week 100
Population: Study Part III analysis set included all participants who were treated with guselkumab during Study Part IIb (Weeks 32 to 64 of the Study, and who were withdrawn from study treatment) and entered Study Part III. Missing data imputed using NRI (participants with missing data at Week 64,76,88 and 100 were considered non-responders).
Measure: Number; unit: Percentage of participants
Arm/Group | Part III: Guselkumab (GUS) | Part III: FAE to Guselkumab
Number analyzed (Participants) | 36 | 12
Percentage of participants | 25 | 8.3

39. Secondary Outcome: Part III: Percentage of Participants Who Achieved Ss-IGA Score of Absence of Disease (0) at Week 100 in Participants With Scalp Psoriasis and Ss-IGA Score>=2 (at Least Mild Disease) at Baseline (Week 0)
Description: as for outcome 11
Time Frame: Week 100
Population: Population included Part III analysis set. Missing data imputed using NRI (participants with missing data at Week 64, 76, 88 and 100 were considered non-responders). Here N (number of participants analyzed) signifies number of participants with Scalp psoriasis and ss-IGA score >=2 at Baseline (Week 0).
Measure: Number; unit: Percentage of participants
Arm/Group | Part III: Guselkumab (GUS) | Part III: FAE to Guselkumab
Number analyzed (Participants) | 34 | 12
Percentage of participants | 14.7 | 8.3

40. Secondary Outcome: Part III: Percentage of Participants Who Achieved an Scalp Specific Investigator´s Global Assessment (Ss-IGA) Score of 0 or 1 at Week 100 in Participants With Scalp Psoriasis and an Ss-IGA Score >=2 (at Least Mild Disease) at Baseline (Week 0)
Description: as for outcome 11
Time Frame: Week 100
Population: Population included Part III analysis set. Missing data imputed using NRI (participants with missing data at Week 64,76,88 and 100 were considered non-responders). Here N (number of participants analyzed) signifies number of participants with Scalp Psoriasis and an ss-IGA Score >=2 (at least mild disease) at Baseline (Week 0).
Measure: Number; unit: Percentage of participants
Arm/Group | Part III: Guselkumab (GUS) | Part III: FAE to Guselkumab
Number analyzed (Participants) | 34 | 12
Percentage of participants | 32.4 | 25.0

41. Secondary Outcome: Part III: Change From Baseline (Week 56) in 36-Item Short-Form Health Survey Version 2 (SF-36 V2) Physical Component Summary (PCS) and Mental Component Summary (MCS) Scores at Week 100
Description: SF-36 V2 is a generic 36-item questionnaire measuring health-related quality of life (HRQL) covering 2 summary measures: physical component summary (PCS) and mental component summary (MCS). The SF-36 consists of 8 subscales (physical function, role limitations due to physical problems, pain, general health perception, vitality, social function, role limitations due to emotional problems, and mental health). Participants self-report on items in a subscale that have between 2-6 choices per item using Likert-type responses (e.g. none of the time, some of the time, etc.). Summations of item scores of the same subscale give the subscale scores, which are transformed into a range from 0 to 100; 0 = worst HRQL, 100=best HRQL. Higher scores indicate better health status.
Time Frame: Baseline (Week 56) and Week 100
Population: Part III analysis set included all participants treated with GUS during Part IIb (Weeks 32 to 64, and who were withdrawn from study treatment) and entered Study Part III. Missing data was imputed using LOCF method.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part III: Guselkumab (GUS) | Part III: FAE to Guselkumab
Number analyzed (Participants) | 36 | 12
Units on a scale
  SF-36 PCS scores: Baseline (Week 56) | 57.8 (3.0) | 54.9 (5.5)
  SF-36 PCS scores: Change at Week 100 | -4.3 (6.7) | -3.7 (7.0)
  SF-36 MCS scores: Baseline (Week 56) | 53.4 (6.2) | 44.2 (11.3)
  SF-36 MCS scores: Change at Week 100 | -2.8 (5.9) | -3.1 (5.9)

42. Secondary Outcome: Part I/IIa: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) (up to Week 32) as a Measure of Safety and Tolerability
Description: An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. Treatment-emergent AEs (TEAEs) were defined as AEs that occurred during active treatment period through Week 32 after the start of initial study drug administration or AEs that were present at Baseline but worsened in severity after the start of initial study drug administration. Safety reported collectively for Part I and Part IIa (that is from Week 0 to Week 32) per planned analysis.
Time Frame: Up to Week 32
Population: Safety analysis set included all participants randomized to 1 of 2 treatment groups (GUS or FAE) at Week 0 and received at least 1 dose of study drug as per actual treatment received during study irrespective of treatment assigned at randomization. Here N (number of subjects analyzed) signifies number of participants evaluable for this OM.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part I/IIa: Guselkumab (GUS) | Part I/IIa: FAE
Number analyzed (Participants) | 60 | 58
Percentage of Participants | 78.3 | 98.3

43. Secondary Outcome: Part IIb: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) (Week 32 to Week 64) as a Measure of Safety and Tolerability
Description: An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs were defined as those AEs that occurred during the active treatment period from Week 32 to Week 56 or the safety follow-up period from Week 56 through Week 64 or those AEs that were present before Week 32 but worsened in severity after Week 32.
Time Frame: Week 32 to Week 64
Population: Study Part IIb analysis set included all participants who entered Study Part IIb and were treated with one of the two treatments (GUS or FAE) at least once during the treatment period from Week 32 to Week 56. Here, n (number of participants analyzed) signifies number of participants analyzed for this OM for specified category.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part IIb: Guselkumab (GUS) | Part IIb: Fumaric Acid Esters (FAE)
Number analyzed (Participants) | 55 | 34
Percentage of Participants
  PASI75 Responders: number analyzed (Participants) | 54 | 14
  PASI75 Responders | 79.6 | 92.9
  PASI75 Non-responders: number analyzed (Participants) | 1 | 20
  PASI75 Non-responders | 0 | 70.0

44. Secondary Outcome: Part III: Percentage of Participants With Adverse Drug Reactions (ADRs) as a Measure of Safety and Tolerability
Description: ADRs were defined as those adverse events with causality 'very likely', 'probable', or 'possible' that occurred during the follow-up extension period from Week 64 to Week 100 or those present before Week 64 but ongoing at Week 64.
Time Frame: Week 64 to Week 100
Population: Study Part III analysis set included all participants who were treated with guselkumab during Study Part IIb (Weeks 32 to 64 of the Study) and entered Study Part III.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part III: Guselkumab (GUS) | Part III: FAE to Guselkumab
Number analyzed (Participants) | 36 | 12
Percentage of Participants | 5.6 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 100
Description: Population included safety analysis set, Part IIb and Part III analysis set. AEs/SAEs till Week 64, and ADRs and deaths from Week 64 to 100 were analyzed and reported. Safety reported collectively for Part I and Part IIa (that is from Week 0 to Week 32) per planned analysis.
Groups:
- Part I/IIa (Week 0 to Week 32): Guselkumab (GUS): In Part I, participants received GUS 100 mg treatment administered as 100 mg/mL solution SC at Weeks 0, 4, 12 and 20. Participants who completed treatment phase until Week 24 entered Part II of study. Participants who completed Part I continued to receive GUS 100 mg SC at Week 28 and 32 during study Part IIa. For participants who discontinued study, a safety follow-up was done at Week 32 (Part I) or 12 weeks after last treatment (whatever came first). For all participants who continued study, safety was followed-up at every visit.
- Part I/IIa (Week 0 to Week 32): Fumaric Acid Esters (FAE): In Part I, Participants received FAE initial/FAE tablets by self-administration at Week 0. The doses were up-titrated and had to be taken every day with different daily doses depending on the optimal individual benefit risk ratio (maximum 6*120 mg/day) according to local prescribing information up to Week 24. Participants who completed the treatment phase until Week 24 entered the Part II of the study. Participants who completed Part I and consented for Part IIa continued to receive commercially available FAE tablets specifically labeled for the study from Week 24 through Week 32 during study Part IIa. For participants who discontinued study, a safety follow-up was done at Week 32 (Part I) or 12 weeks after last treatment (whatever came first). For all participants who continued study, safety was followed-up at every visit.
- Part IIb (Week 32 Through Week 56): Guselkumab (GUS): At Week 32 (study Part IIb), PASI 75 response was evaluated and PASI 75 responders and non-responders of guselkumab arm continued to receive guselkumab 100 mg SC every 8 weeks (weeks 36, 44 and 52). Safety follow up was done at Week 64 (Part II). Participants who discontinued at any timepoint were followed up 12 weeks after last treatment dose. For all participants who continued study, safety was followed-up at every visit.
- Part IIb (Week 32 Through Week 56): Fumaric Acid Esters (FAE): At Week 32, PASI 75 response was evaluated and PASI 75 responders of the FAE arm continued to receive commercially available FAE tablets specifically labeled for the study during Part IIb up to Week 56. Safety follow up was done at Week 64 (Part II). Participants who discontinued at any timepoint were followed up 12 weeks after last treatment dose. For all participants who continued study, safety was followed-up at every visit.
- Part IIb (Week 32 Through Week 56): FAE to Guselkumab: At Week 32, PASI 75 response was evaluated and PASI 75 non-responders of FAE arm were switched to 100 mg guselkumab SC at Weeks 32 and continued at Week 36, 44 and Week 52. Safety follow up was done at Week 64 (Part II). Participants who discontinued at any timepoint were followed up 12 weeks after last treatment dose. For all participants who continued study, safety was followed-up at every visit.
- Part III (Week 64 Through Week 100): Guselkumab: Participants who received guselkumab in Study Part II (participants who started guselkumab treatment at Week 0), had no psoriatic arthritis at baseline and achieved a PASI 90 response at end of Study Part II (Week 56) entered follow-up extension at Week 64 in Study Part III (GUS withdrawal phase) and were followed-up until loss of response or until Week 100.
- Part III (Week 64 Through Week 100): FAE to Guselkumab: At Week 32, PASI 75 response was evaluated and PASI 75 non-responders of FAE arm were switched to GUS and received GUS 100 mg SC at week 32, 36, 44 and 52. Safety follow-up was done at Week 64 (Part II). Participants who discontinued at any timepoint were followed-up 12 weeks after last treatment dose. Participants who switched from FAE to GUS treatment at Week 32, had no psoriatic arthritis at baseline and achieved a PASI 90 response at end of Study Part II (Week 56) entered follow-up extension at Week 64 in Study Part III (GUS withdrawal phase) and were followed-up until loss of response or until Week 100.
Arm/Group | Part I/IIa (Week 0 to Week 32): Guselkumab (GUS) | Part I/IIa (Week 0 to Week 32): Fumaric Acid Esters (FAE) | Part IIb (Week 32 Through Week 56): Guselkumab (GUS) | Part IIb (Week 32 Through Week 56): Fumaric Acid Esters (FAE) | Part IIb (Week 32 Through Week 56): FAE to Guselkumab | Part III (Week 64 Through Week 100): Guselkumab | Part III (Week 64 Through Week 100): FAE to Guselkumab
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/58 | 0/55 | 0/14 | 0/20 | 0/36 | 0/12
Serious Adverse Events (participants affected / at risk) | 3/60 | 2/58 | 3/55 | 1/14 | 2/20 | 0/36 | 0/12
Other Adverse Events (participants affected / at risk) | 47/60 | 57/58 | 43/55 | 13/14 | 14/20 | 2/36 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part I/IIa (Week 0 to Week 32): Guselkumab (GUS) (N=60) | Part I/IIa (Week 0 to Week 32): Fumaric Acid Esters (FAE) (N=58) | Part IIb (Week 32 Through Week 56): Guselkumab (GUS) (N=55) | Part IIb (Week 32 Through Week 56): Fumaric Acid Esters (FAE) (N=14) | Part IIb (Week 32 Through Week 56): FAE to Guselkumab (N=20) | Part III (Week 64 Through Week 100): Guselkumab (N=36) | Part III (Week 64 Through Week 100): FAE to Guselkumab (N=12)
Thymus Enlargement (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part I/IIa (Week 0 to Week 32): Guselkumab (GUS) (N=60) | Part I/IIa (Week 0 to Week 32): Fumaric Acid Esters (FAE) (N=58) | Part IIb (Week 32 Through Week 56): Guselkumab (GUS) (N=55) | Part IIb (Week 32 Through Week 56): Fumaric Acid Esters (FAE) (N=14) | Part IIb (Week 32 Through Week 56): FAE to Guselkumab (N=20) | Part III (Week 64 Through Week 100): Guselkumab (N=36) | Part III (Week 64 Through Week 100): FAE to Guselkumab (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 5 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 21 | 0 | 5 | 1 | 0 | 0
Monocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Middle Ear Inflammation (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Dry Eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Visual Acuity Reduced (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual Impairment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 9 | 0 | 0 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 18 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Defaecation Urgency (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 34 | 0 | 0 | 0 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Faeces Soft (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 6 | 0 | 0 | 0 | 0 | 0
Tooth Disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 5 | 0 | 0 | 1 | 0 | 0
Feeling Hot (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection Site Rash (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Seasonal Allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 5 | 1 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 2 | 1 | 0 | 0 | 1 | 0 | 0
Ear Infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 2 | 1 | 0 | 0 | 0 | 0
Gastrointestinal Infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 2 | 1 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 25 | 19 | 28 | 8 | 8 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Oral Herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Otitis Media (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 2 | 1 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 5 | 0 | 2 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 0 | 0
Skin Candida (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tinea Pedis (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 3 | 1 | 2 | 0 | 0 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bone Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 1 | 0 | 0
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post-Traumatic Neck Syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Traumatic Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 4 | 3 | 3 | 0 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 2 | 1 | 0 | 0 | 1 | 0
Blood Glucose Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Hepatic Enzyme Increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Human Chorionic Gonadotropin Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymph Node Palpable (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases Increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Weight Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Food Intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 2 | 0 | 1 | 0 | 0
Articular Calcification (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3 | 1 | 0 | 0 | 0
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 0 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Giant Cell Tumour of Tendon Sheath (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Carpal Tunnel Syndrome (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 9 | 8 | 3 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Device Breakage (Product Issues) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mood Altered (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 1 | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 0
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Polymorphic Light Eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 5 | 2 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 6 | 0 | 1 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dental Operation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin Neoplasm Excision (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aortic Elongation (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 19 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 4 | 2 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye Haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypothermia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic Steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis Viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis Norovirus (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis Salmonella (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulpitis Dental (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Root Canal Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rotavirus Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood Glucose Decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breath Sounds Abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte Count Increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Lymphocyte Morphology Abnormal (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Protein Urine Present (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
White Blood Cells Urine Positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Femoroacetabular Impingement (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysplastic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Cervicogenic Vertigo (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ketonuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral Venous Disease (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
In Part III, small groups with less subjects generated through Part IIb, and further decline in subjects enrolled in Part III (ie, subjects started guselkumab (GUS) at Week 0/ switched from FAE to GUS in Week 32, and had PASI 90 response at Week 56).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT02951533/Prot_002.pdf
  • Statistical Analysis Plan (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/33/NCT02951533/SAP_003.pdf